CLINICAL TRIAL: NCT06330610
Title: Evaluation de l'efficacité du Support Nutritionnel entéral Intermittent Sur la défaillance d'Organes de Patients de réanimation Sous Ventilation assistée ENteral NUTrition - Continue Intermittent
Brief Title: Evaluation of the Efficiency of Intermittent Enteral Nutrition on Multi-organ Failure From Patients With Mechanical Ventilation in Intensive Care Unit
Acronym: ENNUT-CI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Collaborators: University Hospital, Lille (Other); University Hospital, Caen (Other); Amiens University Hospital (Other); Centre Hospitalier Saint-Philibert, GHICL (Unknown); Centre Hospitalier Intercommunal Elbeuf-Louviers-Val de Reuil (Other Government); Groupe Hospitalier du Havre (Other); Centre Hospitalier de Dieppe (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021/0378/HP
Record Dates: First submitted 2024-03-01; First posted 2024-03-26 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Intermittent Fasting; Septic Shock; Organ Failure, Multiple
Keywords: Enteral nutrition; Mechanical ventilation; Intermittent fasting; Sepsis shock; Organ failure
MeSH Terms: conditions — Intermittent Fasting; Shock, Septic; Multiple Organ Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent enteral nutrition (Experimental): patients that receive intermittent enteral nutrition.
  Interventions: Other: Intermittent enteral nutrition
- continuous enteral nutrition (No Intervention): patients that receive continuous enteral nutrition

INTERVENTIONS:
Other: Intermittent enteral nutrition — Patients will receive intermittent enteral nutrition, defined as 3 60-minute administrations every 8 hours.
  Arms: Intermittent enteral nutrition

SUMMARY:
This study aims to evaluate the efficiency of intermittent enteral nutrition versus continuous enteral nutrition to prevent from organ failures for patients at the acute phase of sepsis shock with mechanical ventilation in ICU.

DETAILED DESCRIPTION:
Some pre-clinical and observational studies have suggested that intermittent fasting may have a positive impact on patients in ICU by increasing protein synthesis, sensibility to insulin, cetogenesis, autophagy by respecting the circadian rhythm. This study aims to evaluate the impact on organ failures of an intermittent enteral nutrition versus continuous enteral nutrition in patients at the acute phase of sepsis shock with mechanical ventilation in the ICU.

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted in ICU for less than 48h, with invasive mechanical ventilation predicted for at least 48h, that can undergo nasogastric feeding for 7 days.
* Patient under vasopressive drugs
* Adult patients (age ≥ 18 years)
* Informed person who has read and signed their consent

  * If the patient is unable to sign their consent (emergency situation), the consent will be signed by a trusted person or a family member, and consent to continue the study will be requested subsequently.
  * If the patient is unable to sign their consent (emergency situation) and no trusted person is present, the patient may be included in the study. In this case, consent to continue the study will be requested from a trusted person as soon as possible, or from the patient if they are able to understand and sign the consent.
* Affiliation to a social security scheme
* No current pregnancy: for women of childbearing age, a beta-HCG blood pregnancy test will be performed upon inclusion; for postmenopausal women, a confirmatory diagnosis must be obtained.

Exclusion Criteria:

* Contraindication to enteral nutrition and/or nasogastric tube insertion: esophageal varices and occlusive syndrome
* Artificial enteral nutrition that cannot be initiated within 48 hours of intubation
* Enteral nutrition ongoing for more than one hour at the time of inclusion
* Need for exclusive or supplemental parenteral nutrition
* Moribund patient
* Person deprived of liberty by an administrative or judicial decision or person placed under judicial protection/guardianship or curatorship
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2024-07-09 (Actual); Primary Completion 2027-10-09 (Estimated); Study Completion 2027-10-09 (Estimated)

PRIMARY OUTCOMES:
Evolution of variation of the SOFA (Sepsis-related organ failure assessment) score. | day-1 (nutrition start) and day-7
  Comparison of variation of the SOFA score between patients with intermittent nutrition versus patients with continuous nutrition.

SECONDARY OUTCOMES:
evaluation of caloric intake | from day-1 (nutrition start) to day-7
  evaluation of caloric intake (kcal/day)
evaluation of protein intake | from day-1 (nutrition start) to day-7
  evaluation of protein intake (g/kg/day)
Measurement of nutritionnal status | day-1 (nutrition start) and day-7
  measurement of weight (kg)
Evaluation of the digestive tolerance | from day-1 (nutrition start) to day-7
  Number of vomit (number)
Evaluation of the nosocomial infections | from day-1 (nutrition start) to day-7
  Type of infection
Adverse events | from day-1 (nutrition start) to day-7
  Number of adverse event
Evaluation of the metabolic response | day 1, day 4 and day 7
  metabolomics analysis (96 proteins assay)
Evaluation of the duration of hospitalisation | day 1 to day 90
  number of days at hospital
Evaluation of the intensive care neuromuscular weakness | Up to day 10
  MRC score
Evaluation of death | from day 1 to day 90
  Death data collection
Evaluation of quality of life | up to day 90
  SF-36 score

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Rouen, Rouen, France, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Atherton PJ, Etheridge T, Watt PW, Wilkinson D, Selby A, Rankin D, Smith K, Rennie MJ. Muscle full effect after oral protein: time-dependent concordance and discordance between human muscle protein synthesis and mTORC1 signaling. Am J Clin Nutr. 2010 Nov;92(5):1080-8. doi: 10.3945/ajcn.2010.29819. Epub 2010 Sep 15. PMID 20844073
- [Background] McNelly AS, Bear DE, Connolly BA, Arbane G, Allum L, Tarbhai A, Cooper JA, Hopkins PA, Wise MP, Brealey D, Rooney K, Cupitt J, Carr B, Koelfat K, Damink SO, Atherton PJ, Hart N, Montgomery HE, Puthucheary ZA. Effect of Intermittent or Continuous Feed on Muscle Wasting in Critical Illness: A Phase 2 Clinical Trial. Chest. 2020 Jul;158(1):183-194. doi: 10.1016/j.chest.2020.03.045. Epub 2020 Apr 2. PMID 32247714
- [Background] Gonzalez JT, Dirks ML, Holwerda AM, Kouw IWK, van Loon LJC. Intermittent versus continuous enteral nutrition attenuates increases in insulin and leptin during short-term bed rest. Eur J Appl Physiol. 2020 Sep;120(9):2083-2094. doi: 10.1007/s00421-020-04431-4. Epub 2020 Jul 10. PMID 32651634
- [Background] Marcheva B, Ramsey KM, Peek CB, Affinati A, Maury E, Bass J. Circadian clocks and metabolism. Handb Exp Pharmacol. 2013;(217):127-55. doi: 10.1007/978-3-642-25950-0_6. PMID 23604478
- [Background] Baggs JE, Hogenesch JB. Genomics and systems approaches in the mammalian circadian clock. Curr Opin Genet Dev. 2010 Dec;20(6):581-7. doi: 10.1016/j.gde.2010.08.009. PMID 20926286
- [Background] Jamshed H, Beyl RA, Della Manna DL, Yang ES, Ravussin E, Peterson CM. Early Time-Restricted Feeding Improves 24-Hour Glucose Levels and Affects Markers of the Circadian Clock, Aging, and Autophagy in Humans. Nutrients. 2019 May 30;11(6):1234. doi: 10.3390/nu11061234. PMID 31151228
- [Background] Pickel L, Sung HK. Feeding Rhythms and the Circadian Regulation of Metabolism. Front Nutr. 2020 Apr 17;7:39. doi: 10.3389/fnut.2020.00039. eCollection 2020. PMID 32363197
- [Background] Gunst J. Recovery from critical illness-induced organ failure: the role of autophagy. Crit Care. 2017 Aug 7;21(1):209. doi: 10.1186/s13054-017-1786-y. PMID 28784175
- [Background] Vanhorebeek I, Gunst J, Derde S, Derese I, Boussemaere M, Guiza F, Martinet W, Timmermans JP, D'Hoore A, Wouters PJ, Van den Berghe G. Insufficient activation of autophagy allows cellular damage to accumulate in critically ill patients. J Clin Endocrinol Metab. 2011 Apr;96(4):E633-45. doi: 10.1210/jc.2010-2563. Epub 2011 Jan 26. PMID 21270330
- [Background] Hermans G, Casaer MP, Clerckx B, Guiza F, Vanhullebusch T, Derde S, Meersseman P, Derese I, Mesotten D, Wouters PJ, Van Cromphaut S, Debaveye Y, Gosselink R, Gunst J, Wilmer A, Van den Berghe G, Vanhorebeek I. Effect of tolerating macronutrient deficit on the development of intensive-care unit acquired weakness: a subanalysis of the EPaNIC trial. Lancet Respir Med. 2013 Oct;1(8):621-629. doi: 10.1016/S2213-2600(13)70183-8. Epub 2013 Sep 10. PMID 24461665
- [Background] Martinez-Lopez N, Tarabra E, Toledo M, Garcia-Macia M, Sahu S, Coletto L, Batista-Gonzalez A, Barzilai N, Pessin JE, Schwartz GJ, Kersten S, Singh R. System-wide Benefits of Intermeal Fasting by Autophagy. Cell Metab. 2017 Dec 5;26(6):856-871.e5. doi: 10.1016/j.cmet.2017.09.020. Epub 2017 Oct 26. PMID 29107505
- [Background] Newman JC, Verdin E. beta-Hydroxybutyrate: A Signaling Metabolite. Annu Rev Nutr. 2017 Aug 21;37:51-76. doi: 10.1146/annurev-nutr-071816-064916. PMID 28826372
- [Background] Cox PJ, Kirk T, Ashmore T, Willerton K, Evans R, Smith A, Murray AJ, Stubbs B, West J, McLure SW, King MT, Dodd MS, Holloway C, Neubauer S, Drawer S, Veech RL, Griffin JL, Clarke K. Nutritional Ketosis Alters Fuel Preference and Thereby Endurance Performance in Athletes. Cell Metab. 2016 Aug 9;24(2):256-68. doi: 10.1016/j.cmet.2016.07.010. Epub 2016 Jul 27. PMID 27475046
- [Background] Zou X, Meng J, Li L, Han W, Li C, Zhong R, Miao X, Cai J, Zhang Y, Zhu D. Acetoacetate Accelerates Muscle Regeneration and Ameliorates Muscular Dystrophy in Mice. J Biol Chem. 2016 Jan 29;291(5):2181-95. doi: 10.1074/jbc.M115.676510. Epub 2015 Dec 8. PMID 26645687
- [Background] Goossens C, Weckx R, Derde S, Dufour T, Vander Perre S, Pauwels L, Thiessen SE, Van Veldhoven PP, Van den Berghe G, Langouche L. Adipose tissue protects against sepsis-induced muscle weakness in mice: from lipolysis to ketones. Crit Care. 2019 Jul 1;23(1):236. doi: 10.1186/s13054-019-2506-6. PMID 31262340
- [Background] Stekovic S, Hofer SJ, Tripolt N, Aon MA, Royer P, Pein L, Stadler JT, Pendl T, Prietl B, Url J, Schroeder S, Tadic J, Eisenberg T, Magnes C, Stumpe M, Zuegner E, Bordag N, Riedl R, Schmidt A, Kolesnik E, Verheyen N, Springer A, Madl T, Sinner F, de Cabo R, Kroemer G, Obermayer-Pietsch B, Dengjel J, Sourij H, Pieber TR, Madeo F. Alternate Day Fasting Improves Physiological and Molecular Markers of Aging in Healthy, Non-obese Humans. Cell Metab. 2019 Sep 3;30(3):462-476.e6. doi: 10.1016/j.cmet.2019.07.016. Epub 2019 Aug 27. PMID 31471173
- [Background] de Cabo R, Mattson MP. Effects of Intermittent Fasting on Health, Aging, and Disease. N Engl J Med. 2019 Dec 26;381(26):2541-2551. doi: 10.1056/NEJMra1905136. No abstract available. PMID 31881139
- [Background] Thiessen SE, Van den Berghe G, Vanhorebeek I. Mitochondrial and endoplasmic reticulum dysfunction and related defense mechanisms in critical illness-induced multiple organ failure. Biochim Biophys Acta Mol Basis Dis. 2017 Oct;1863(10 Pt B):2534-2545. doi: 10.1016/j.bbadis.2017.02.015. Epub 2017 Feb 17. PMID 28219766
- [Background] Van Dyck L, Casaer MP. Intermittent or continuous feeding: any difference during the first week? Curr Opin Crit Care. 2019 Aug;25(4):356-362. doi: 10.1097/MCC.0000000000000617. PMID 31107308
- [Background] Deane AM, Chapman MJ, Reintam Blaser A, McClave SA, Emmanuel A. Pathophysiology and Treatment of Gastrointestinal Motility Disorders in the Acutely Ill. Nutr Clin Pract. 2019 Feb;34(1):23-36. doi: 10.1002/ncp.10199. Epub 2018 Oct 7. PMID 30294835
- [Background] Van Dyck L, Vanhorebeek I, Wilmer A, Schrijvers A, Derese I, Mebis L, Wouters PJ, Van den Berghe G, Gunst J, Casaer MP. Towards a fasting-mimicking diet for critically ill patients: the pilot randomized crossover ICU-FM-1 study. Crit Care. 2020 May 24;24(1):249. doi: 10.1186/s13054-020-02987-3. PMID 32448392
- [Background] Singer P, Blaser AR, Berger MM, Alhazzani W, Calder PC, Casaer MP, Hiesmayr M, Mayer K, Montejo JC, Pichard C, Preiser JC, van Zanten ARH, Oczkowski S, Szczeklik W, Bischoff SC. ESPEN guideline on clinical nutrition in the intensive care unit. Clin Nutr. 2019 Feb;38(1):48-79. doi: 10.1016/j.clnu.2018.08.037. Epub 2018 Sep 29. PMID 30348463
- [Derived] Tebani A, Demailly Z, Bekri S, Maizel J, Marchalot A, Bourel C, Du Cheyron D, Michot JB, Schnell G, Vanderlinden T, Tamion F. Clinical and metabolic phenotyping of continuous versus intermittent ENteral NUTrition in ventilated adults with shock: ENNUT trial protocol. BMJ Open. 2025 Aug 1;15(7):e099761. doi: 10.1136/bmjopen-2025-099761. PMID 40750277